CLINICAL TRIAL: NCT02808351
Title: Multicenter Randomized Controlled Study of Berberine for Prevention of Contrast-Induced Acute Kidney Injury in Patients With Diabetes and Renal Insufficient
Brief Title: Berberine Prevent Contrast-induced Nephropathy in Patients With Diabetes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Shaoliang Chen, MD, Director of Cardiology and Cath Lab, Vice President of Nanjing First Hospital, Nanjing First Hospital, Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NFH20160611
Record Dates: First submitted 2016-06-12; First posted 2016-06-21 (Estimated); Last update posted 2022-03-29 (Actual); Status verified 2022-03

CONDITIONS: Diabetes Mellitus; Chronic Kidney Disease
MeSH Terms: conditions — Diabetes Mellitus; Renal Insufficiency, Chronic | interventions — Berberine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Berberine (Experimental): Preoperative berberine 300 mg administration for at least 6 hours before interventional procedure, post-procedure berberine administration 100 mg at 24, 48 hours after procedure.
  Interventions: Drug: Berberine
- Blank control (No Intervention): Blank control of berberine administration

INTERVENTIONS:
Drug: Berberine
  Arms: Berberine

SUMMARY:
The number of cardiac angiography and percutaneous coronary interventions (PCI) has increased steadily in recent years. This has resulted in the increasing incidence of contrast-induced nephropathy (CIN). Major risk factors for CIN include older age, diabetes mellitus (DM), chronic kidney disease(CKD), the concurrent use of nephrotoxic drugs, hemodynamic instability, etc. Importantly, DM appears to act as a risk multiplier, meaning that in a patient with CKD it amplifies the risk of CIAKI.

The aim of this multicenter prospective, randomized, controlled study is to evaluate whether berberine treatment during and after the perioperative period would reduce the risk of CIN in a high-risk population of patients with both DM and CKD undergoing coronary angiography or noncoronary angiography, and the influence of such potential benefit on short-term outcome.

ELIGIBILITY:
Inclusion Criteria:

* Planned diagnostic coronary or peripheral artery angiography
* Type 2 diabetes mellitus
* CKD stages ≥2
* Statin naive, or not on statin treatment for at least 14 days
* Withdrawal metformin or aminophylline for 48h before angiography
* Total iodixanol volume

Exclusion Criteria:

* Hypersensitivity to iodine-containing compounds and berberine
* Ketoacidosis
* Lactic acidosis
* CKD stages 1, 5 (eGFR≥90ml/min per 1.73m2 or eGFR<15ml/min per 1.73m2)
* STEMI
* NYHA class IV or hemodynamic instability
* Administration of any iodinated contrast medium within 14 days before randomization
* LDL-C<1.82mmol/L（70mg/dL）
* Hepatic dysfunction (ALT 3 times greater than upper normal limit)
* Thyreoid insufficiency
* Renal artery Stenosis(unilateral >70％ or bilateral stenosis>50％)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2021-12 (Actual); Study Completion 2021-12 (Actual)

PRIMARY OUTCOMES:
Contrast-induced nephropathy | 72 hours
  An absolute increase in serum creatinine (SCr) >=0.5mg/dL（>=44.2μmmol/L）or a >= 25% increase in SCr from baseline to 72 hours after the procedure

SECONDARY OUTCOMES:
Major adverse renal events | 30 days
  The composite of hospitalization for aggravated renal function, acute renal failure, dialysis or hemofiltration, aggravated at least 1 class of heart function, acute left ventricular failure or death from all causes.

CONTACTS AND LOCATIONS:
Overall Officials: Shaoliang Chen, Study Chair — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- Nanjing First Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No